CLINICAL TRIAL: NCT02855710
Title: Rhythm Game Park: a Training of the Rhythmic Skills With a Serious Game to Improve Gait and Cognitive Abilities in Parkinson's Disease
Brief Title: A Training of the Rhythmic Skills With a Serious Game to Improve Gait and Cognitive Abilities in Parkinson's Disease
Acronym: RGP
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: end of inclusion period
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Laboratory Parole et Langage UMR 7309 (Unknown); Laboratory EUROMOV EA 2991 (Unknown); Université Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9499
Record Dates: First submitted 2016-07-27; First posted 2016-08-04 (Estimated); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- No training (Other): Parkinsonian Patients with no Rhythm Workers training perceptive timing and senrorimotor timing
  Interventions: Other: No Rhythm workers training
- Perceptive timing training (Other): Parkinsonian Patients with Rhythm Workers training perceptive timing
  Interventions: Other: Rhythm workers training Perceptive timing
- Sensorimotor timing training (Other): Parkinsonian Patients with Rhythm Workers training sensorimotor timing
  Interventions: Other: Rhythm workers training sensorimotor timing
- Healthy volunteers (Other): Healthy people with Rhythm Workers training perceptive timing
  Interventions: Other: Rhythm workers training Perceptive timing

INTERVENTIONS:
Other: Rhythm workers training Perceptive timing — Perceptive timing training
  Arms: Healthy volunteers; Perceptive timing training
Other: Rhythm workers training sensorimotor timing — Sensorimotor timing training
  Arms: Sensorimotor timing training
Other: No Rhythm workers training — No training
  Arms: No training

SUMMARY:
This project aims at assessing the opposite relation, namely the effect of a training of the general timing abilities on gait in Parkinson's disease. Timing rehabilitation will be done by the means of a serious game. Serious games are more and more used to improve the compliance and the efficacy of reeducaiton programs. Overall, we propose to test a low-cost tool for rehabilitation.

DETAILED DESCRIPTION:
Auditory rythmic cueing is a method consisting in presenting a regular auditory stimulus (metronom or music) when someone is walking. It is known to improve gait in pathologies such as Parkinson's disease. It has also an effect on general timing abilities (e.g. tapping the beat of the music). This project aims at assessing the opposite relation, namely the effect of a training of the general timing abilities on gait in Parkinson's disease. Timing rehabilitation will be done by the means of a serious game. Serious games are more and more used to improve the compliance and the efficacy of reeducaiton programs. Overal, we propose to test a low-cost tool for rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* age < 18
* good understanding of the nature, the goal and the methodology of the study
* signing of the informed consent
* being insured with a social security
* Diagnostic of idiopathic Parkinson's disease following the Queen Square Brain Bank (Hughes, 1992)
* Hoehn et Yahr between 2 and 3
* mild to moderate walk and speech deficits (Item MDS-UPDRS)
* stable therapy one month before inclusion for all the duration of the study

Exclusion Criteria:

* Atypic Parkinson Syndrom (oculomotor troubles, early falls, hallucinations, MoCA<20, early dysautonomy)
* dystonia ou dyskinesia preventing from using a tablet (item MDS-UPDRS4.2 >2)
* Unable to move without help (walking stick, walker, wheelchair) (item MDS-UPDRS 2.12 >2)
* adult protected by law
* deprivation of liberty
* High propability of non compliance to the protocol
* pregnant women, nursing women
* moderate to severe auditory trouble
* Severe walk fluctuations item MDS-UPDRS 4.4 >2)
* Pacemaker or neurosensorial device or heart defebrillator
* Cochlear implants
* ferromagnetic external bodies claose to the brain
* Metallic prothesis
* agitated, non cooperative patient
* claustrophobic patient
* neuro-surgical shunt valves
* dental appliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Rythmic capacities | 3 months
  Evaluate the effect of the training of the rythmic capacities (Sensorimotor timing abilities) on the walk and the speak

SECONDARY OUTCOMES:
cognitive functions | 3 months
  Evaluate the cognitive functions by Neurospsychologic tests
Mesure of the neural reorganisation | 3 months
  Evaluate the structure et connectivity by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Christian Gény, MD, Study Chair — University Hospital, Montpellier
Locations (1):
- Gui de Chauliac Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No